CLINICAL TRIAL: NCT03307707
Title: Heart Failure and Early Stage Chronic Kidney Disease -Mineral Bone Disorder : the Importance of the New Biomarkers
Brief Title: New Heart Failure Biomarkers in Early Stage Chronic Kidney Disease-Mineral and Bone Disorder
Acronym: CKD-MBD-HF
Status: Completed | Type: Observational
Sponsor: Pr. Semir Nouira (Other)
Responsible Party: Sponsor-Investigator, Pr. Semir Nouira, Professor, University of Monastir
Organization: University of Monastir (Other)
Other Study IDs: CKD-MBD-HF
Record Dates: First submitted 2017-10-04; First posted 2017-10-12 (Actual); Last update posted 2017-10-12 (Actual); Status verified 2017-10

CONDITIONS: Kidney Disease, Chronic; Heart Failure
Keywords: FGF23; klotho; Mineral Bone Disorder
MeSH Terms: conditions — Renal Insufficiency, Chronic; Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples were centrifuged, the plasma were collected and stored at -80°C until utilization.

GROUPS / COHORTS (2):
- Heart Failure (HF): subjects with a Left Ventricular Ejection Fraction (LVEF) <50% or LVEF >50% and E/e'>10.
- No Heart Failure (NHF): subjects with LVEF>50%

SUMMARY:
the objective of this study is to :

-Determinate wether the circulating levels of iFGF23 and klotho can be a predictor biomarker of HF in patients with CKD-MBD.

DETAILED DESCRIPTION:
The disorders of mineral metabolism and bone disease are common complications in CKD patients and they are associated with increased morbidity and mortality.

Abnormalities of the vasculature are seen in early CKD, producing vascular stiffness contributing to left ventricular hypertrophy and its pathophysiology involves newly discovered hormones, such as the fibroblast Growth factor 23 (FGF23) and α- klotho.

The FGF receptor and its co-receptor klotho moderate these effects. FGF23 levels inflate early in in the advancement of CKD stage to attain levels in CKD stage 5D.

But we still have few knoweledges if these markers can have some drawbacks for predicting CVD in early stage CKD.

ELIGIBILITY:
Inclusion Criteria:

* Early CKD stage
* Heart failure

Exclusion Criteria:

* Infections
* cancer
* corticoid therapy
* renal replacement therapy
* Advanced CKD stage

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: subjects who visited the emmergency departement or the nephrology departement , meeting the criteria inclusion and have given a written consent .
Sampling Method: Probability Sample
Enrollment: 111 (Actual)
Dates: Start 2015-06-15 (Actual); Primary Completion 2015-09-30 (Actual); Study Completion 2015-12-30 (Actual)

PRIMARY OUTCOMES:
Fibroblast Growth Factor 23 (FGF23) | completed data base (after 4 months)
  compare the circulating levels of FGF23 (pg/ml) in the two groups .
Alpha Klotho | completed data base (after 4 months)
  compare the circulating levels of klotho (ng/ml) in the two groups .

CONTACTS AND LOCATIONS:
Overall Officials: Lamti Feten, PhD student, Study Chair — Research Laboratory (LR12SP18) University of Monastir Tunisia, Tunisia and Research Unit (UR17ES29) Faculty of Pharmacy , Monastir